CLINICAL TRIAL: NCT04285255
Title: Quality of Recovery of Opioid Free Anaesthesia Versus Opioids Anaesthesia Within Enhanced Recovery Protocol Following Laparoscopic Sleeve Gastrectomy in Saudi Arabia, Randomized Controlled Trial
Brief Title: Quality of Recovery Following Opioids Free Anaesthesia in Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al Mashfa Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OFA
Record Dates: First submitted 2020-02-22; First posted 2020-02-26 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2020-03

CONDITIONS: Narcotics; Recovery Quality; Analgesia; Bariatric Surgery
MeSH Terms: conditions — Agnosia | interventions — Fentanyl; Ketamine; Dexmedetomidine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: only the anaesthetist is one aware of the study groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioids anesthesia (Active Comparator): received propofol-fentanyl induction of anaesthesia plus ultrasound-guided Bilateral oblique subcostal TAP block using 20ml of bupivacaine hydrochloride 0.25% (Marcaine, Astra Zeneca UK) in each side (total volume of 40 ml) deposited equally on each side
  Interventions: Drug: Fentanyl; Procedure: Oblique subcostal transversus abdominis plane block
- OFA (Active Comparator): received preinduction with dexmeditomidine 0.1µg.kg-1 over 10 min. Induction with propofol 1.5 mg.kg-1-ketamine (ketofol 3:1 mixture) induction plus maintenance mixture of dexmedetomidine 0.5µg.kg-1.h-1, ketamine 0.5mg.kg-1.h-1, and lidocaine 1 mg.kg-1.h-1 plus ultrasound-guided Bilateral oblique subcostal TAP block using 20ml of bupivacaine hydrochloride 0.25% (Marcaine, Astra Zeneca UK) in each side (total volume of 40 ml) deposited equally on each side
  Interventions: Drug: Ketamine; Drug: Dexmedetomidine Injection [Precedex]; Procedure: Oblique subcostal transversus abdominis plane block; Drug: Lidocaine

INTERVENTIONS:
Drug: Fentanyl — opioids anaesthesia
  Arms: Opioids anesthesia
Drug: Ketamine — ketamine induction and analgesia as opioids free anaesthesia versus opioids analgesia
  Arms: OFA
Drug: Dexmedetomidine Injection [Precedex] — alpha 2 agonist with sedative, analgesic effect
  Arms: OFA
Procedure: Oblique subcostal transversus abdominis plane block — Bupivacaine 0.25% injected under ultrasound usage in the transversus abdominis plane
Drug: Lidocaine — infusion of lidocaine 2%(1mg/kg/h)
  Arms: OFA

SUMMARY:
Laparoscopic sleeve gastrectomy is widely employed nowadays. Multimodal analgesia approach is implemented within the enhanced recovery protocol in our facility to improve participants' recovery. Due to side effects of narcotics, the may adversely affect the quality of recovery, the investigators intended to test the efficacy of opioids free anaesthesia on the quality of recovery and postoperative narcotic use.

ELIGIBILITY:
Inclusion Criteria:

* 70 ASA II - III adult patients (18-60 years old)
* Elective laparoscopic bariatric surgery.
* Body mass index (BMI) is from 40 to 60
* Trocar sites at or above the umbilicus (T 10 dermatome).

Exclusion Criteria:

* Allergy to amino-amide local anaesthetics,
* presence of coagulopathy
* local skin infection at injection sites,
* preoperative chronic dependence upon opioid and NSAID medications,
* liver or renal insufficiency,
* history of psychiatric or neurological disease, deafness,
* previous open surgery,
* patients who need to be converted to open surgery with more tissue trauma,
* ASA (American society of anesthesiologists) class above III were excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Quality of recovery 40 questionnaire (QoR-40) | At 6 hours
  postoperative quality of recovery
Quality of recovery 40 questionnaire (QoR-40) | At 24th h (period of time between 6 and 24 hours) as repeated measurement
  postoperative quality of recovery

SECONDARY OUTCOMES:
Pethidine consumption | 24 hours
Numerical rating scale (NRS) | 24 hours
  visual analogue scale postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Al Mashfa medical center, Khobar, Eastern Provence, Saudi Arabia

REFERENCES:
- [Derived] Ibrahim M, Elnabtity AM, Hegab A, Alnujaidi OA, El Sanea O. Combined opioid free and loco-regional anaesthesia enhances the quality of recovery in sleeve gastrectomy done under ERAS protocol: a randomized controlled trial. BMC Anesthesiol. 2022 Jan 21;22(1):29. doi: 10.1186/s12871-021-01561-w. PMID 35062872